CLINICAL TRIAL: NCT04490564
Title: A Clinical Performance Study to Validate the Use of Novel Molecular Diagnostic Assays for the Detection of Cancer Biomarkers in Peripheral Blood and Primary Tumor Tissue of Patients With Recurrent/Metastatic HNSCC, NSCLC or Melanoma.
Brief Title: Validation of Molecular Diagnostic Assays to Detect Cancer Biomarkers in Blood and Primary Tumor in HNSCC/NSCLC/Melanoma
Status: Completed | Type: Observational
Sponsor: Pharmassist Ltd (Industry)
Collaborators: University of Athens (Other)
Responsible Party: Sponsor
Other Study IDs: CBS-PD-L1a
Record Dates: First submitted 2020-02-20; First posted 2020-07-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Non Small Cell Lung Cancer; Melanoma
Keywords: Liquid biopsy; CTC; PD-L1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Melanoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CTCs of peripheral blood and primary tumor tissue (FFPEs) samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HNSCC, NSCLC, melanoma Patients: The study population are subjects with a confirmed diagnosis of recurrent or metastatic head and neck squamous cell carcinoma (HNSCC), who are going to receive PD-1 inhibitor nivolumab or ii) metastatic Non-Small Cell Lung Cancer (NSCLC), who are going to receive PD-1 inhibitor, e.g. nivolumab, pembrolizumab or iii) metastatic melanoma, who are going to receive PD-1 inhibitor, e.g. nivolumab, embrolizumab. The selected inclusion/exclusion criteria have been set to include in the performance study appropriate population of interest, as broad as possible, but to exclude these subjects that have another current malignancy or any history of recent malignancy within 3 years.
  Interventions: Diagnostic Test: PD-L1 Kit
- Healthy volunteers: In case of healhty volunteers, only peripheral blood samples will be collected.
  Interventions: Diagnostic Test: PD-L1 Kit

INTERVENTIONS:
Diagnostic Test: PD-L1 Kit — Clinical performance of PD-L1 kit in CTCs of peripheral blood and tumor tissue samples

SUMMARY:
Conventional biopsy and surgical tumor resection are invasive procedures that capture only one instance of the progression of the tumor. However, the genome of tumor is not static, but it is constantly altered during treatment.

Liquid biopsy is a non-invasive approach based on the extraction of information through peripheral blood analysis. It makes it possible to characterize the development of a solid tumor in real time, through detailed molecular analysis of circulating genetic material in peripheral blood.

DETAILED DESCRIPTION:
Conventional biopsy and surgical tumor resection are invasive procedures that capture only one instance of the progression of the tumor. However, the genome of tumor is not static, but it is constantly altered during treatment.

Liquid biopsy is a non-invasive approach based on the extraction of information through peripheral blood analysis. It makes it possible to characterize the development of a solid tumor in real time, through detailed molecular analysis of circulating genetic material in peripheral blood.

Study procedure:

1. Initial Visit (V0-Baseline): For the purposes of the study the following information will be collected: the demographics, medical and social history, the characteristics of the disease (stage, molecular characterization e.t.c) and the treatment regimen that is followed. As part of the visit, 20 mL of peripheral blood will be drawn prior to their treatment according to physician's suggestion as per common clinical practice. Blood samples will be then sent to ACTC laboratory for plasma/CTC isolation, DNA and RNA extraction and subsequent test for biomarkers. Primary tumor tissue samples will be also collected.
2. Follow-up visit (V1): All patients will provide a 10 mL peripheral blood sample during their planned visit at the end of a series of immunotherapy cycles as per clinical practice and physician's judgment. More specifically:

   For HNSCC/NSCLC: at the end of four (4) treatment cycles with nivolumab (2 months) or at the end of three (3) treatment cycles with pembrolizumab (2 months) or on disease progress (PD) For melanoma: at 6 months after treatment initiation (antiPD-1) Blood samples will be then sent to laboratory for plasma/CTC isolation, DNA and RNA extraction and subsequent test for biomarkers. Clinical response (CR, PR, SD, PD) will be also documented.
3. Follow-up visit (V2): All patients will provide a 10 mL peripheral blood sample on progress of the disease or at the end of the observation period, as diagnosed during their planned visit as per clinical practice and physician's judgment. Blood samples will be then sent to laboratory

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 18 years of age.
2. Patients with a diagnosis of

   1. recurrent or metastatic head and neck squamous cell carcinoma (HNSCC), who are going to receive PD-1 inhibitor nivolumab OR
   2. metastatic Non-Small Cell Lung Cancer (NSCLC), who are going to receive PD-1 inhibitor, e.g. nivolumab, pembrolizumab,OR
   3. metastatic melanoma, who are going to receive to receive PD-1 inhibitor, e.g. nivolumab, pembrolizumab.
3. Available tumor tissue sample for immunohistochemical and molecular analysis.
4. Life expectancy ≥ 4 months.
5. Signed informed consent form.

Exclusion Criteria:

1. Male or female younger than 18 years old.
2. History of another malignancy within 3 years or current 2nd primary malignancy.
3. Patients that have not signed the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 155 subjects as follows: 25 patients with metastatic/recurrent HNSCC 120 patients with metastatic NSCLC 10 patients with metastatic melanoma 30 healthy subjects
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Clinical performance of PD-L1 kit in CTCs of peripheral blood and tumor tissue samples | 12 months
  The performance of PD-L1 kit at baseline in CTCs (using IF as reference method) and tumor tissue samples (using IHC as reference method) will be assessed via Sensitivity, Specificity, Positive and Negative Predictive Values, Positive and Negative Likelihood Ratios, Accuracy and Diagnostic Odds Ratio.

SECONDARY OUTCOMES:
To study correlations between PD-L1 expression in serial liquid samples with patients' responsiveness to therapy. | 18 months
  1. Clinical response to the selected treatment (CR, PR, SD, PD)
  2. Survival status

OTHER OUTCOMES:
To study mutation status of BRAF gene in tumor tissue samples and blood samples (CTC, plasma ctDNA) of metastatic melanoma patients | 18 months
  Mutation profile of BRAF in CTCs, plasma-ctDNA and tumor tissues of metastatic melanoma patients will be evaluated using PCR-molecular assays
To study the presence of biomarkers in tumor tissue and blood liquid biopsy samples (at baseline). | 18 months
  Molecular profile of cancer biomarkers in tumor tissue and peripheral blood samples will be evaluated using PCR-molecular assays

CONTACTS AND LOCATIONS:
Locations (6):
- Greece (6):
  - University General Hospital of Alexandroupoli, Alexandroupoli, Alexandroupolis
  - Sotiria Thoracic Diseases Hospital of Athens, Athens, Attica
  - Aretaieio University Hospital of Athens, Athens, Attica
  - University General Hospital of Athens Attikon, Athens, Attica
  - Metropolital Hospital, Piraeus, Piraeus
  - Bioclinic, Thessaloniki, Thessaloniki